CLINICAL TRIAL: NCT01318980
Title: A Single Dose, Crossover Study in Healthy Female Subjects to Assess the Regional Absorption and Bioavailability of 100 mg GSK2190915A
Brief Title: A Single Dose Study to Assess the Regional Absorption and Bioavailability of 100mg GSK2190915A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 114604
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: ADME; IV radiolabelled; pharmacokinetics
MeSH Terms: conditions — Asthma | interventions — 3-(3-tert-butylsulfanyl-1-(4-(6-ethoxypyridin-3-yl)benzyl)-5-(5-methylpyridin-2-ylmethoxy)-1H-indol-2-yl)-2,2-dimethylpropionic acid; Tablets, Enteric-Coated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Period 1 Cohort 1 - GSK2190915 100mg (Experimental): Period 1 - GSK2190915 100mg tablet.
  Interventions: Drug: GSK2190915 100mg milled tablet
- Period 1 Cohort 2 - GSK2190915 100mg plus microtracer (Experimental): Period 1 - GSK2190915 100mg tablet plus [14C] radiolabelled GSK2190915 microtracer solution.
  Interventions: Drug: GSK2190915 100mg milled tablet; Drug: [14C] radiolabelled GSK2190915 solution
- Period 2 GSK2190915 100mg to proximal small bowel (Experimental): 100mg of ground half 200mg GSK2190915 tablet administered to the proximal small bowel via Enterion capsule.
  Interventions: Drug: GSK2190915 100mg milled tablet administered to the proximal small bowel.
- Period 3 GSK2190915 100 mg to distal small bowel (Experimental): 100mg of ground half 200mg GSK2190915 tablet administered to the distal small bowel via Enterion capsule.
  Interventions: Drug: GSK2190915 100mg milled tablet administered to the distal small bowel.
- Period 4 - GSK 100mg enteric-coated tablet (Experimental): 100mg enteric-coated GSK2190915 coated tablet.
  Interventions: Drug: GSK2190915 100mg enteric-coated tablet.

INTERVENTIONS:
Drug: GSK2190915 100mg milled tablet — Taken orally
  Arms: Period 1 Cohort 1 - GSK2190915 100mg; Period 1 Cohort 2 - GSK2190915 100mg plus microtracer
Drug: [14C] radiolabelled GSK2190915 solution — Microtracer solution
  Arms: Period 1 Cohort 2 - GSK2190915 100mg plus microtracer
Drug: GSK2190915 100mg milled tablet administered to the proximal small bowel. — Ground half of a 200mg tablet. Administered via Enterion capsule.
  Arms: Period 2 GSK2190915 100mg to proximal small bowel
Drug: GSK2190915 100mg milled tablet administered to the distal small bowel. — Ground half of a 200mg tablet. Administered via Enterion capsule.
  Arms: Period 3 GSK2190915 100 mg to distal small bowel
Drug: GSK2190915 100mg enteric-coated tablet. — Taken orally
  Arms: Period 4 - GSK 100mg enteric-coated tablet

SUMMARY:
GSK2190915 is a high affinity 5-lipoxygenase-activating protein (FLAP) inhibitor that attenuates the production of leukotrienes through the blockage of the first step in the leukotriene pathway, 5-lipoxygenase (5-LO) activation. GSK2190915 inhibits the production of leukotriene B4 (LTB4) and cysteinyl leukotrienes (cysLTs).

This is an open label, 4-way, 4-treatment period, non-randomised, crossover study with an interim analysis. The GSK2190915 formulations used in this study will be: a 100mg and 200mg milled tablet, a 100mg enteric-coated tablet, and a [14C] radiolabelled GSK2190915 intravenous solution.

This study aims to determine the pharmacokinetics and absolute bioavailability of GSK2190915 to enable optimisation of suitable formulations to be used in clinical development Fourteen subjects will be dosed to ensure data in 10 at the end of the clinical study. Seven of the subjects will receive an IV microtracer in addition to the other treatments.

DETAILED DESCRIPTION:
GSK2190915 is a high affinity 5-lipoxygenase-activating protein (FLAP) inhibitor that attenuates the production of leukotrienes through the blockage of the first step in the leukotriene pathway, 5-lipoxygenase (5-LO) activation. Leukotrienes are potent inflammatory molecules produced mainly by mast cells, eosinophils, monocytes/macrophage and neutrophils in response to allergic or inflammatory stimuli. GSK2190915 inhibits the production of leukotriene B4 (LTB4) and cysteinyl leukotrienes (cysLTs).

This is an open label, 4-way, 4 treatment period, non-randomised, single-dose crossover study with an interim analysis following the third treatment period. The GSK2190915 formulations used are: milled 100mg and 200mg tablets, a 100mg enteric-coated tablet, and a [14C] radiolabelled GSK2190915 intravenous solution.

There will be 4 periods. Period 1 includes two cohorts (of 7 subjects each), both of which will be administered the 100mg GSK2190915 milled tablet orally; however, the second cohort will in addition be dosed with an intravenous radiolabelled infusion of the drug. In the second period, a 100mg dose of milled GSK2190915 tablet (a ground half of a 200mg tablet) is administered directly to the proximal small bowel using an Enterion capsule. The same dose is repeated in the third period, but is administered directly to the distal small bowel. An interim analysis will then follow. The decision to proceed will be made following a review of the pharmacokinetic data from the first three treatments. In the fourth and final period, the treatment will be a 100mg enteric-coated tablet of GSK2190915 administered orally. There will be a minimum washout of 7 days in between each period.

This study aims to determine the pharmacokinetics and absolute bioavailability of GSK2190915 to enable optimisation of suitable formulations to be used in clinical development. Periods 1 to 3 will characterise the absolute bioavailability of GSK2190915 using IV tracer and oral formulation, in addition to defining the regional absorption characteristics of the drug when released in the proximal and distal parts of the gastro-intestinal tract. The fourth period will investigate the oral bioavailability of an enteric coated formulation of GSK2190915.

Fourteen subjects will be dosed to ensure data in 10 at the end of the clinical study. Seven of the subjects (in cohort 2, Period 1) will receive an IV microtracer in addition to the other treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females as determined by an experienced study physician, based on a medical evaluation including medical history, physical examination, neurological examination, laboratory tests and electrocardiogram (ECG). A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures;
* Females must be either:
* Of non-childbearing potential, defined as pre-menopausal females with a documented tubal ligation or hysterectomy or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. [Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 9.4 of the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.]
* Of child-bearing potential and agrees to use one of the contraception methods listed in Section 9.4 of the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 3 months after the last dose.
* Aged 18-65 years;
* Body Mass Index (BMI) of 18-35 kilogram per sqare metre (km/m2);
* Subjects must demonstrate their ability to swallow an empty size 000 capsule;
* Must be willing and able to participate in the whole study and must provide written informed consent;
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase and bilirubin ≤ 1.5xUpper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%);
* QTcB or QTcF < 450 msec
* Subjects of child-bearing potential must agree to use one of the contraception methods listed in Section 9.4 from the time of the first dose of study medication until 3 months following the last dose.
* Exclusion Criteria:
* Participation in a clinical research study involving investigational drugs or dosage forms within the previous 3 months or 4 months if new chemical entity (NCE);
* Subjects who have previously been enrolled in this study;
* Subjects who have ever sought advice from or been referred to a General Practitioner or counsellor for abuse or misuse of alcohol, non medical drugs, medicinal drugs or other substance abuse e.g. solvents;
* Subjects who admit to any current or previous use of Class A drugs such as opiates, cocaine, ecstasy, lysergic acid diethylamide (LSD) and intravenous amphetamines (Subjects who admit to occasional past use of cannabis will not be excluded as long as they have a negative drugs of abuse test and have been abstinent for at least 12 months;)
* Positive drugs of abuse test result;
* Regular alcohol consumption >14 units per week (1 Unit = ½ pint beer, a 25 milliLitre (mL) shot of 40% spirit or a 125 mL glass of wine);
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening;
* Radiation exposure from clinical trials, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 milliSieverts (mSv) in the last twelve months or 10 mSv in the last five years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study;
* Subjects must not have had any 14C exposure within the last 12 months.
* Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the Principal Investigator (PI);
* History of gastrointestinal surgery (with the exception of appendectomy unless it was performed within the previous 12 months);
* History of clinically significant cardiovascular, renal, hepatic, respiratory and particularly gastrointestinal disease, especially peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's Disease or Irritable Bowel Syndrome;
* History of adverse reaction or allergy to study drug or its excipients, e.g. lactose or rescue medication (if specified by the Sponsor);
* If subject suffers from hayfever they must not have or be expecting to have symptoms during the study period;
* Acute diarrhoea or constipation in the 7 days before the predicted first study day. If screening occurs >7 days before the first study day, this criterion will be determined on first study day. Diarrhoea will be defined as the passage of liquid faeces and/or a stool frequency of greater than three times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day;
* Donation, or significant loss as judged by the investigator, of blood within the previous three months;
* Presence of non-removable metal objects such as metal plates, screws, etc, in the abdominal region of the body (with the exception of sterilisation clips);
* Subjects will be excluded from the study if they are considered by the PI to be at risk of transmitting, through blood or other body fluids, the agents responsible for acquired immunodeficiency syndrome (AIDS) or other sexually transmitted disease or hepatitis;
* Positive Hepatitis B Virus, Hepatitis C Virus or Human Immunodeficiency Virus (HIV)results;
* Unwillingness or inability to follow the procedures outlined in the protocol;
* Subject is mentally or legally incapacitated;
* Failure to satisfy the PI of fitness to participate for any other reason.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-09-30 (Actual); Primary Completion 2011-03-11 (Actual); Study Completion 2011-03-11 (Actual)

PRIMARY OUTCOMES:
Characterisation of the maximum concentration (Cmax), the time of Cmax (tmax) and Area Under the plasma concentration-time Curve (AUC) for intravenous and oral pharmacokinetics | 1 month
Determination of AUC data for all routes of administration to permit calculation of relative and absolute bioavailability where appropriate. | 1 month
Assessment of regiospecific bioavailability of GSK2190915A based on tmax, Cmax, and AUC to assist in subsequent oral formulation/delivery options for GSK2190915A | 1 month

SECONDARY OUTCOMES:
To collect further information about the safety and tolerability of GSK2190915A by assessing: physical examination, safety laboratory tests, vital signs, electrocardiogram (ECG), adverse events. | 1 month
Quantitative and cumulative recovery of radiocarbon in urine and faeces to permit an assessment of deposition route for intravenous GSK2190915A. | 1 month
Collection of bile to allow profiling of metabolites of GSK2190915A. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114604 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114604?search=study&study_ids=114604#rs
- Available data/document: Annotated Case Report Form: 114604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114604 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register